CLINICAL TRIAL: NCT05820165
Title: Study on Brain Structure and Function Imaging in Patients With Cerebral Venous Outflow Disturbance
Brief Title: Brain Imaging in Cerebral Venous Outflow Disturbance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Other Study IDs: COVD-BI
Record Dates: First submitted 2023-04-14; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Abnormal Cerebral Venous Sinus Morphology; Internal Jugular Vein Stenosis; Image
MeSH Terms: interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood samples from enrolled participants are drawn by nurse using containing coagulant tubes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CVOD-WS: Cerebral Venous Outflow Disturbance with symptoms such as tinnitus cerebri，somnipathy ，anxiety ，depression and cognitive decline
  Interventions: Radiation: high-resolution 3D-T1; Radiation: diffusion tensor imaging (DTI); Radiation: resting-state functional magnetic resonance imaging (rs-fMRI); Radiation: arterial spin labeling (ASL) perfusion magnetic resonance imaging (MRI); Radiation: susceptibility-weighted images (SWIs)
- CVOD-WOS: Cerebral Venous Outflow Disturbance without symptoms such as tinnitus cerebri，somnipathy ，anxiety ，depression and cognitive decline
  Interventions: Radiation: high-resolution 3D-T1; Radiation: diffusion tensor imaging (DTI); Radiation: resting-state functional magnetic resonance imaging (rs-fMRI); Radiation: arterial spin labeling (ASL) perfusion magnetic resonance imaging (MRI); Radiation: susceptibility-weighted images (SWIs)
- HC: Healthy control
  Interventions: Radiation: high-resolution 3D-T1; Radiation: diffusion tensor imaging (DTI); Radiation: resting-state functional magnetic resonance imaging (rs-fMRI); Radiation: arterial spin labeling (ASL) perfusion magnetic resonance imaging (MRI); Radiation: susceptibility-weighted images (SWIs)

INTERVENTIONS:
Radiation: high-resolution 3D-T1 — Subjects undergo a high-resolution 3D-T1 imaging to obtain structural images
Radiation: diffusion tensor imaging (DTI) — Subjects undergo a DTI imaging to obtain images of white matter lesions
Radiation: resting-state functional magnetic resonance imaging (rs-fMRI) — Subjects undergo rs-fMRI to investigate the differences in intra-regional brain activity and inter-regional functional connectivity
Radiation: arterial spin labeling (ASL) perfusion magnetic resonance imaging (MRI) — Subjects undergo arterial spin labeling (ASL) perfusion magnetic resonance imaging (MRI) to clarify the difference of cerebral blood flow (CBF) perfusion in certain regions
Radiation: susceptibility-weighted images (SWIs) — Subjects undergo susceptibility-weighted images (SWIs) to segment the vein network

SUMMARY:
Cerebral venous outflow disturbance can lead to cerebral hemodynamic disturbances, altered cerebrospinal fluid dynamics, cerebral venous blood stasis, increased cerebral venous pressure and decreased cerebral perfusion, cerebral white matter sparing-like changes, and widening of retinal vessel diameter. These changes are associated with numerous neurological signs and symptoms. Therefore, understanding the brain structural and functional changes in patients with cerebral venous outflow disturbance is essential to provide specific imaging evaluation indicators and new diagnosis and treatment methods for patients with cerebral venous return disorders.

DETAILED DESCRIPTION:
Cerebral venous outflow disturbance can lead to cerebral hemodynamic disturbances, altered cerebrospinal fluid dynamics, cerebral venous blood stasis, increased cerebral venous pressure and decreased cerebral perfusion, cerebral white matter sparing-like changes, and widening of retinal vessel diameter. These changes are associated with numerous neurological signs and symptoms. A number of central nervous system disorders such as transient global amnesia, transient monocular blindness, primary labor headaches, and even Parkinson's have been reported to be closely associated with internal jugular vein stenosis. Other common clinical manifestations include sleep disturbances, tinnitus, tinnitus, headache, visual impairment, optic papilledema, hearing loss, cognitive decline and neck discomfort and even autonomic dysfunction. The main objective of this study is to investigate the structural and functional network changes in patients with cerebral venous outflow disturbance using different brain imaging techniques, to clarify the correlation between symptoms of cerebral venous outflow disturbance and brain structure and function; to identify areas with corresponding structural and functional changes in patients with cerebral venous outflow disturbance and or comorbid symptoms, and to provide specific imaging assessment indicators and new diagnostic and treatment tools for patients with cerebral venous outflow disturbance and comorbid symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral venous outflow disturbance( moderate to severe stenosis in cerebral venous sinus or intracranial jugular veins ) is confirmed by two of magnetic resonance venography (MRV), computed tomography venography (CTV) or digital subtraction angiography (DSA)
* Accompanying symptoms such as tinnitus cerebri, cognitive decline, anxiety depression, sleep disorders, etc. for more than 6 months

Exclusion Criteria:

* ear primary disease medicine related intracranial hypertension; Systemic disease of abnormal metabolism or inflammation; moderate to severe stenosis in intracranial, carotid or vertebral arteries; intracranial lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with cerebral venous outflow disturbance( moderate to severe stenosis in cerebral venous sinus or intracranial jugular veins )
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
voxel-based morphometry | at admission
  Voxel-based morphometry (VBM) is used to obtain the relative gray matter volume (GMV) and WM volume (WMV)

SECONDARY OUTCOMES:
The amplitude of low-frequency fluctuations (ALFF) | at admission
  The amplitude of low-frequency fluctuations (ALFF) is used to investigate the differences in intra-regional brain activity and inter-regional functional connectivity

OTHER OUTCOMES:
Regional homogeneity (ReHo) | at admission
  The Regional homogeneity (ReHo) is used to investigate the differences in intra-regional brain activity and inter-regional functional connectivity
Voxel-wise functional connectivity (FC) | at admission
  The Voxel-wise functional connectivity (FC) is used to investigate the differences in intra-regional brain activity and inter-regional functional connectivity
Tract-based spatial statistics (TBSS) analysis | at admission
  Tract-based spatial statistics (TBSS) analysis is used to investigate fractional anisotropy (FA) values
Mini-Mental State Examination(MMSE) | at admission
  Mini-Mental State Examination(MMSE) is used to evaluate global cognitive function
Montreal Cognitive Assessment (MoCA) | at admission
  Montreal Cognitive Assessment (MoCA) is used to evaluate global cognitive function
Subjective Cognitive Decline（SCD） | at admission
  Subjective Cognitive Decline（SCD）is used to evaluate global cognitive function
Self-Rating Anxiety Scale（SAS） | at admission
  Self-Rating Anxiety Scale（SAS）is used to evaluate neuropsychological change
Self-rating depression scale（SDS） | at admission
  Self-rating depression scale（SDS）is used to evaluate neuropsychological change
Pittsburgh sleep quality index（PSQI） | at admission
  Pittsburgh sleep quality index（PSQI）is used to evaluate somnipathy
Tinnitus handicap inventory（THI） | at admission
  Tinnitus handicap inventory（THI）is used to evaluate tinnitus cerebri

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD.PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu hospital;Capital Medical University, Beijin, XI Cheng District, China

REFERENCES:
- [Background] Luan Y, Wang C, Jiao Y, Tang T, Zhang J, Teng GJ. Prefrontal-Temporal Pathway Mediates the Cross-Modal and Cognitive Reorganization in Sensorineural Hearing Loss With or Without Tinnitus: A Multimodal MRI Study. Front Neurosci. 2019 Mar 12;13:222. doi: 10.3389/fnins.2019.00222. eCollection 2019. PMID 30930739